CLINICAL TRIAL: NCT01667536
Title: A Phase 2 Assessment of the Diagnostic Accuracy of 99mTc-MIP-1404 Imaging in Men With High-Risk Prostate Cancer Scheduled for Radical Prostatectomy (RP) and Extended Pelvic Lymph Node Dissection (EPLND) Compared to Histopathology
Brief Title: A Phase 2 Study With MIP-1404 in Men With High-Risk PC Scheduled for RP and EPLND Compared to Histopathology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIP-1404-201
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Cancer
Keywords: PROSTATE CANCER; HIGH-RISK; PROSTATECTOMY SURGERY; NEWLY DIAGNOSED
MeSH Terms: conditions — Prostatic Neoplasms | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: 99mTc-MIP-1404 (Experimental): 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404
  Interventions: Drug: Drug: 99mTc-MIP-1404

INTERVENTIONS:
Drug: Drug: 99mTc-MIP-1404 — A single dose of 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404
  Other Names: MIP-1404

SUMMARY:
This was a multicenter, multi-reader, open-label, Phase 2 study assessing the safety and performance characteristics of MIP 1404 imaging in the detection of prostate gland and pelvic lymph node cancer. Comparative performance characteristics between MIP 1404 imaging and MRI were also assessed, as judged by histopathology results.

DETAILED DESCRIPTION:
This is a single arm, open label study of approximately 100 high-risk prostate cancer patients scheduled for prostatectomy and extended pelvic lymph node dissection. Patients receive a single IV dose of 99mTc-MIP-1404 (study drug) followed by SPECT/CT scan 3-6 hours after injection. As standard of care, patients will undergo prostatectomy and extended pelvic lymph node dissection (EPLND) within three weeks of study drug dosing. 99mTc-MIP-1404 image data will be evaluated for visible uptake and compared with histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older.
* Ability to provide signed informed consent and willingness to comply with protocol requirements.
* Biopsy confirmed presence of adenocarcinoma of the prostate gland.
* At high-risk for metastatic disease by a stage of cT3, cT4, or a total nomogram score of greater than or equal to 130.
* Scheduled to undergo radical prostatectomy with extended pelvic lymph node dissection.
* Agree to use an acceptable form of birth control for a period of 7 days after the 99mTc MIP-1404 injection.

Exclusion Criteria:

* Participating would significantly delay the scheduled standard of care therapy.
* Administered a radioisotope within 5 physical half lives prior to study drug injection.
* Have any medical condition or other circumstances that, in the opinion of the investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study.
* Have a contraindication for MR imaging.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scherr, M.D., Principal Investigator — New York Presbyterian Hospital-Cornell; Jeffrey Karnes, MD, Principal Investigator — Mayo Clinic; Kevin Slawin, MD, Principal Investigator — University of Texas Vanguard Urologic Research Foundation; Thomas Keane, MD, Principal Investigator — Medical University of South Carolina; Edouard Trabulsi, MD, Principal Investigator — Thomas Jefferson University / Jefferson Urology Associates; David Jarrard, MD, Principal Investigator — University of Wisconsin, Madison; William Ellis, MD, Principal Investigator — University of Washington; Judd Moul, MD, Principal Investigator — Duke University; Eric Klein, MD, Principal Investigator — Glickman Urology & Kidney Institute, Cleveland Clinic; Bertram Yuh, MD, Principal Investigator — City of Hope National Cancer Center; Steven Joniau, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Alberto Briganti, MD, Principal Investigator — Vita-Salute University San Raffaele; Paolo Gontero, MD, Principal Investigator — University of Turin, Italy; Mikhail I Shkolnik, MD, Principal Investigator — Federal State Public Institution Russian Research center for Radiology and Surgical Technologies under the Federal agency for High-tech medical care; Petr A Karlov, MD, Principal Investigator — St. Petersburg State Public Medical Institution: "Clinical Oncological Center"; Vsevolod B Matveev, MD, Principal Investigator — Federal Public State Institution "Russian Oncology Research Center n.a. N.N. Blokhin under the Russian Academy of medical sciences"; Boris Ya Alexeev, MD, Principal Investigator — Moscow Oncology Research Institute n.a. P.A. Hertsen; Sergey V Mishugin, MD, Principal Investigator — City Clinical Hospital # 57; Oleg B Karyakin, Principal Investigator — Federal State Public Institution "Medical Radiology Research Center" of Healthcare Ministry and Social Development of Russian Federation; Alexander K Nosov, MD, Principal Investigator — Research Institute of Oncology n.a. Professor N.N. Petrov under the Federal Agency for Healthcare and Social Development; Sergey B Petrov, MD, Principal Investigator — All-Russia Centre for Urgent Care and Radiation Medicine named after A.M. Nikiforov under the Ministry of the Russian Federation for Civil Defence, Emergencies and Elimination of Consequences of Natural Disasters; Milan Hora, MD, PhD, Principal Investigator — University Hospital Plzen, Department of Urology; Josef Stolz, MD, Principal Investigator — University Hospital Motol, Clinic of Urology; Vladimir Student, MD, PhD, Principal Investigator — University Hospital Olomouc, Clinic of Urology; Marek Krolupper, MD, Principal Investigator — Hospital Na Bulovce, Department of Urology; Michael Pesl,, MD, Principal Investigator — General University Hospital in Prague, Clinic of Urology; Roman Zachoval,, MD, PhD, MBA, Principal Investigator — Thomayer's Hospital; Marcin Matuszewski, MD, PhD, Principal Investigator — University Clinical Centre, Department of Urology; Henryk Zielinski, MD, Principal Investigator — University Hospital Plzen, Department of Urology; Jerzy Sokolowski, MD, PhD, Principal Investigator — Provincial Specialist Hospital in Wroclaw, Department of Urology; Tomasz Szydelko, MD, PhD, Principal Investigator — 4th Military Teaching Hospital and Polyclinic,; Geza Boszormenyi-Nagy, MD, Principal Investigator — Bajcsy-Zsilinszky Hospital, Department of Urology; Peter Tenke, MD, Principal Investigator — Jahn Ferenc South Pest Hospital, Department of Urology; Istvan Buzogany, MD, Principal Investigator — Peterfy Sandor Street Hospital, Department of Urology; Michiel Sedelaar, MD, Principal Investigator — UMC St. Radboud Nijmegen
Locations (35):
- United States (10):
  - City of Hope National Cancer Center, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Hospital - Cornell, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Glickman Urology & Kidney Institute, Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University / Jefferson Urology Associates, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Vanguard Urologic Research Foundation, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- University Hospitals Leuven, Leuven, Belgium
- Czechia (6):
  - University Hospital Olomouc, Clinic of Urology, Olomouc
  - University Hospital Plzen, Department of Urology, Pilsen
  - General University Hospital in Prague, Clinic of Urology, Prague
  - Thomayer's Hospital, Prague
  - University Hospital Motol, Clinic of Urology, Prague
  - Hospital Na Bulovce, Department of Urology, Prague
- Hungary (3):
  - Bajcsy-Zsilinszky Hospital, Department of Urology, Budapest
  - Peterfy Sandor Street Hospital, Department of Urology, Budapest
  - Jahn Ferenc South Pest Hospital, Department of Urology, Budapest
- Italy (2):
  - Vita-Salute University San Raffaele, Milan
  - University of Turin, Torino
- UMC St. Radboud Nijmegen, Nijmegen, Netherlands
- Poland (4):
  - University Clinical Centre, Department of Urology, Gdansk
  - University Hospital Plzen, Department of Urology, Warsaw
  - 4th Military Teaching Hospital and Polyclinic,, Wroclaw
  - "Provincial Specialist Hospital in Wroclaw, Department of Urology, Wroclaw
- Russia (8):
  - City Clinical Hospital # 57, Moscow
  - Federal Public State Institution "Russian Oncology Research Center n.a. N.N. Blokhin under the Russian Academy of medical sciences", Moscow
  - Moscow Oncology Research Institute n.a. P.A. Hertsen, Moscow
  - Federal State Public Institution "Medical Radiology Research Center" of Healthcare Ministry and Social Development of Russian Federation, Obninsk
  - All-Russia Centre for Urgent Care and Radiation Medicine named after A.M. Nikiforov under the Ministry of the Russian Federation for Civil Defence, Emergencies and Elimination of Consequences of Natural Disasters, Saint Petersburg
  - Federal State Public Institution Russian Research center for Radiology and Surgical Technologies under the Federal agency for High-tech medical care, Saint Petersburg
  - Research Institute of Oncology n.a. Professor N.N. Petrov under the Federal Agency for Healthcare and Social Development, Saint Petersburg
  - St. Petersburg State Public Medical Institution: "Clinical Oncological Center", Saint Petersburg

REFERENCES:
- [Background] American Cancer Society, Inc., Surveillance Research; Cancer Facts & Figures, 2012
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Hovels AM, Heesakkers RA, Adang EM, Jager GJ, Strum S, Hoogeveen YL, Severens JL, Barentsz JO. The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis. Clin Radiol. 2008 Apr;63(4):387-95. doi: 10.1016/j.crad.2007.05.022. Epub 2008 Feb 4. PMID 18325358
- [Background] Pinto JT, Suffoletto BP, Berzin TM, Qiao CH, Lin S, Tong WP, May F, Mukherjee B, Heston WD. Prostate-specific membrane antigen: a novel folate hydrolase in human prostatic carcinoma cells. Clin Cancer Res. 1996 Sep;2(9):1445-51. PMID 9816319
- [Background] Smith-Jones PM, Vallabahajosula S, Goldsmith SJ, Navarro V, Hunter CJ, Bastidas D, Bander NH. In vitro characterization of radiolabeled monoclonal antibodies specific for the extracellular domain of prostate-specific membrane antigen. Cancer Res. 2000 Sep 15;60(18):5237-43. PMID 11016653
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Murphy GP, Elgamal AA, Su SL, Bostwick DG, Holmes EH. Current evaluation of the tissue localization and diagnostic utility of prostate specific membrane antigen. Cancer. 1998 Dec 1;83(11):2259-69. PMID 9840525
- [Background] Ghosh A, Heston WD. Tumor target prostate specific membrane antigen (PSMA) and its regulation in prostate cancer. J Cell Biochem. 2004 Feb 15;91(3):528-39. doi: 10.1002/jcb.10661. PMID 14755683
- [Background] Perner S, Hofer MD, Kim R, Shah RB, Li H, Moller P, Hautmann RE, Gschwend JE, Kuefer R, Rubin MA. Prostate-specific membrane antigen expression as a predictor of prostate cancer progression. Hum Pathol. 2007 May;38(5):696-701. doi: 10.1016/j.humpath.2006.11.012. Epub 2007 Feb 22. PMID 17320151
- [Background] Silver DA, Pellicer I, Fair WR, Heston WD, Cordon-Cardo C. Prostate-specific membrane antigen expression in normal and malignant human tissues. Clin Cancer Res. 1997 Jan;3(1):81-5. PMID 9815541
- [Background] Luthi-Carter R, Barczak AK, Speno H, Coyle JT. Molecular characterization of human brain N-acetylated alpha-linked acidic dipeptidase (NAALADase). J Pharmacol Exp Ther. 1998 Aug;286(2):1020-5. PMID 9694964
- [Background] Troyer JK, Beckett ML, Wright GL Jr. Detection and characterization of the prostate-specific membrane antigen (PSMA) in tissue extracts and body fluids. Int J Cancer. 1995 Sep 4;62(5):552-8. doi: 10.1002/ijc.2910620511. PMID 7665226
- [Background] Chang SS, Reuter VE, Heston WD, Bander NH, Grauer LS, Gaudin PB. Five different anti-prostate-specific membrane antigen (PSMA) antibodies confirm PSMA expression in tumor-associated neovasculature. Cancer Res. 1999 Jul 1;59(13):3192-8. PMID 10397265
- [Background] Maresca KP, Hillier SM, Femia FJ, Keith D, Barone C, Joyal JL, Zimmerman CN, Kozikowski AP, Barrett JA, Eckelman WC, Babich JW. A series of halogenated heterodimeric inhibitors of prostate specific membrane antigen (PSMA) as radiolabeled probes for targeting prostate cancer. J Med Chem. 2009 Jan 22;52(2):347-57. doi: 10.1021/jm800994j. PMID 19111054
- [Background] Hillier SM, Maresca KP, Femia FJ, Marquis JC, Foss CA, Nguyen N, Zimmerman CN, Barrett JA, Eckelman WC, Pomper MG, Joyal JL, Babich JW. Preclinical evaluation of novel glutamate-urea-lysine analogues that target prostate-specific membrane antigen as molecular imaging pharmaceuticals for prostate cancer. Cancer Res. 2009 Sep 1;69(17):6932-40. doi: 10.1158/0008-5472.CAN-09-1682. Epub 2009 Aug 25. PMID 19706750
- [Background] Godoy G, Chong KT, Cronin A, Vickers A, Laudone V, Touijer K, Guillonneau B, Eastham JA, Scardino PT, Coleman JA. Extent of pelvic lymph node dissection and the impact of standard template dissection on nomogram prediction of lymph node involvement. Eur Urol. 2011 Aug;60(2):195-201. doi: 10.1016/j.eururo.2011.01.016. Epub 2011 Jan 18. PMID 21257258
- [Background] Rao JN, Scott AJ. A simple method for the analysis of clustered binary data. Biometrics. 1992 Jun;48(2):577-85. PMID 1637980
- [Background] Durkalski VL, Palesch YY, Lipsitz SR, Rust PF. Analysis of clustered matched-pair data for a non-inferiority study design. Stat Med. 2003 Jan 30;22(2):279-90. doi: 10.1002/sim.1385. PMID 12520562
- [Derived] Hillier SM, Maresca KP, Lu G, Merkin RD, Marquis JC, Zimmerman CN, Eckelman WC, Joyal JL, Babich JW. 99mTc-labeled small-molecule inhibitors of prostate-specific membrane antigen for molecular imaging of prostate cancer. J Nucl Med. 2013 Aug;54(8):1369-76. doi: 10.2967/jnumed.112.116624. Epub 2013 Jun 3. PMID 23733925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: 99mTc-MIP-1404
Started | 105
Completed | 105 (105 subjects comprised the safety popn, defined as all subjects who received an MIP-1404 injection.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug: 99mTc-MIP-1404
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 105

OUTCOME MEASURES:

1. Primary Outcome: Assess the Ability of 99mTc-MIP-1404 to Detect Prostate Cancer Within the Prostate Gland.
Description: For the prostate gland, sensitivity values refer to the number of subjects in the study, i.e., the percentages of true positive subjects correctly identified by the imaging technique. Pathology results were used as the truth standard for all imaging analyses.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: The primary analysis population is defined as all subjects who completed prostate and lymph node SPECT/CT MIP-1404 imaging, underwent EPLND, and had histopathology results. This population is one less than the safety population (n=105)
Measure: Number (90% Confidence Interval); unit: % sensitivity
Arm/Group | Drug: 99mTc-MIP-1404
Number analyzed (Participants) | 104
% sensitivity | 94.2 [89.2 to 97.0]

2. Secondary Outcome: Assess the Ability of MIP-1404 to Detect Metastatic Prostate Cancer Within Pelvic Lymph Nodes
Description: For lymph nodes, sensitivity values refer to the number of subjects in the study, i.e., the percentages of true positive subjects correctly identified by the imaging technique. Pathology results were used as the truth standard for all imaging analyses.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: The primary analysis population, defined as all subjects who completed prostate and lymph node SPECT/CT MIP-1404 imaging, underwent EPLND, and had histopathology results, was used for this endpoint. A total of 3025 nodes were removed from 103 subjects (mean 29.6, range 1-88). Of these, 79 nodes were positive by pathology in 33 subjects.
Measure: Number (90% Confidence Interval); unit: % sensitivity
Arm/Group | Drug: 99mTc-MIP-1404
Number analyzed (Participants) | 33
% sensitivity | 33.3 [19.8 to 46.9]

3. Secondary Outcome: Assess the Ability of MIP-1404 to Detect the Extent and Location of Prostate Cancer Within the Prostate Gland
Description: For specific segments of the prostate, a sensitivity value refers to the number of evaluable segments (histologically examined "tissue-segments") from all subjects, i.e., the percentages of true positive segments correctly identified by the imaging technique.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: % sensitivity
Units Other Than Participants: Prostate Segments
Groups:
- Drug: 99mTc-MIP-1404: 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404 Drug: 99mTc-MIP-1404: A single dose of 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404
Arm/Group | Drug: 99mTc-MIP-1404
Number analyzed (Participants) | 104
Number analyzed (Prostate Segments) | 519
% sensitivity | 44.4 [36.1 to 45.0]

4. Secondary Outcome: Assess the Ability of MIP-1404 to Detect the Specific Location of Metastatic Prostate Cancer Within Anatomic Pelvic Lymph Node Regions
Description: For specific segments of the lymph nodes, a sensitivity value refers to the number of evaluable segments (histologically examined "tissue-segments") from all subjects, i.e., the percentages of true positive segments correctly identified by the imaging technique.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: % sensitivity
Units Other Than Participants: Lymph Node Segments
Arm/Group | Drug: 99mTc-MIP-1404
Number analyzed (Participants) | 104
Number analyzed (Lymph Node Segments) | 1144
% sensitivity | 8.1 [3.2 to 19.3]

5. Secondary Outcome: Assess the Comparative Performance of MIP-1404 Against MRI for Detection of Prostate Cancer Within the Prostate Gland.
Description: Comparative performance characteristics between MIP-1404 imaging and MRI were analyzed for the prostate gland. MIP-1404 and MRI sensitivities were derived from case positive histopathology results.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: All subjects who completed prostate SPECT/CT MIP-1404 and MRI imaging and had histopathology results.
Measure: Number; unit: % specificity
Groups:
- Drug: 99mTc-MIP-1404: 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404
  Drug: 99mTc-MIP-1404: A single dose of 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404. Sensitivity based on 99mTc-MIP-1404 imaging.
- Drug: 99mTc-MIP-1404 + MRI: Drug: 99mTc-MIP-1404: A single dose of 20 ±3 mCi intravenous (IV) injection of 99mTc-MIP-1404. Sensitivity based on MRI imaging.
Arm/Group | Drug: 99mTc-MIP-1404 | Drug: 99mTc-MIP-1404 + MRI
Number analyzed (Participants) | 96 | 96
% specificity | 93.8 | 85.4

6. Secondary Outcome: Assess the Comparative Performance of MIP-1404 Against MRI for Detection of Metastatic Prostate Cancer Within Pelvic Lymph Nodes.
Description: Comparative performance characteristics between MIP-1404 imaging and MRI were analyzed for the lymph nodes. MIP-1404 and MRI sensitivities were derived from case positive histopathology results.
Time Frame: Within 3-6 hours of dosing SPECT/CT images will be taken
Population: All subjects who completed lymph node SPECT/CT MIP-1404 and MRI imaging, underwent EPLND, and had histopathology results.
Measure: Number; unit: % sensitivity
Arm/Group | Drug: 99mTc-MIP-1404 | Drug: 99mTc-MIP-1404 + MRI
Number analyzed (Participants) | 33 | 32
% sensitivity | 33.3 | 12.5

ADVERSE EVENTS:
Time Frame: Day 0 (day of dosing) to Day 21 post study drug injection.
Arm/Group | Drug: 99mTc-MIP-1404
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less